CLINICAL TRIAL: NCT03925935
Title: A Phase 1, Open Label, Non-randomized, Multi-Center Trial of AB-205 in Adults With Lymphoma Undergoing High-Dose Therapy and Autologous Stem Cell Transplantation
Brief Title: Trial of AB-205 in Adults With Lymphoma Undergoing High-Dose Therapy and Autologous Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Angiocrine Bioscience (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AB-205-001
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Hodgkin Lymphoma; Non-hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Intervention Model Description: AB-205 dose escalation based on safety.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Up to 3 sequential dose escalation cohorts of AB-205
  Interventions: Biological: AB-205

INTERVENTIONS:
Biological: AB-205 — Engineered human umbilical vein endothelial cells

SUMMARY:
A phase 1, open label, multi-center trial of AB-205 in adults with Hodgkin or non-Hodgkin lymphoma who are in chemo-sensitive remission undergoing high-dose therapy, with or without radiation, and autologous stem cell transplantation (HDT-ASCT). Subjects will receive AB-205 infusion following autologous stem cell transfusion on Day 0.

ELIGIBILITY:
INCLUSION CRITERIA

* Diagnosis of Hodgkin lymphoma (HL) or non-Hodgkin lymphoma (NHL) who are candidates for HDT-ASCT with one of the following conditioning regimens:

  * carmustine, etoposide, cytarabine, melphalan (BEAM)
  * cyclophosphamide, carmustine, etoposide (CBV)
  * thiotepa, busulphan, cyclophosphamide (TBC)
  * additional myeloablative chemotherapy-based conditioning regimens may be permitted with the approval of the medical monitor
* Adjunct radiation therapy to HDT will be allowed.
* Adequate organ function is required, defined as follows:

  * Serum bilirubin ≤ 2 mg/dL, unless benign congenital hyperbilirubinemia
  * AST, ALT, and alkaline phosphatase < 3 times the upper limit of normal
  * Creatinine clearance ≥ 40 ml/min (calculated by Cockcroft Gault)
  * LVEF ≥ 45% by MUGA or resting echocardiogram
  * Pulmonary function (FEV1 and corrected DLCO) ≥ 45% predicted
  * Adequate performance status ECOG ≤1
* For female subjects of childbearing potential:

  * A negative serum or urine pregnancy test at screening.
  * Subject must be willing to use a recommended method of contraception from the start of the screening period and throughout the study period.
* For males who can father a child and are having intercourse with females of childbearing potential who are not using adequate contraception:

  - Subject must be willing to use a recommended method of contraception and refrain from sperm donation from the start of conditioning therapy for at least 1 year after completion and discussion with a treating physician.
* Willingness and ability to comply with scheduled visits, drug administration plan, protocol-specified laboratory tests, other study procedures, and study restrictions.
* Ability to provide written informed consent.

EXCLUSION CRITERIA

* History of prior ASCT.
* Active malignancy other than the one for which the subject is undergoing HDT-ASCT. (Subjects with cervical carcinoma in situ or localized basal or squamous cell carcinoma treated with definitive surgery are eligible.)
* Subjects with a serious concomitant medical condition that could interfere with the conduct of the clinical trial, such as unstable angina, renal failure requiring hemodialysis, or active infection requiring IV antibiotics.
* Active Human Immunodeficiency Virus (HIV) infection and Acquired Immunodeficiency Syndrome (AIDS).
* Females who are pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 30 days or longer after chemotherapy treatment discontinuation if required by prescribing information for chemotherapy agents received during the study.
* Subjects who have known hypersensitivity reactions to bovine (cow) proteins or documented allergy to DMSO.
* Subject has other conditions that in the opinion of the investigator would place the subject at increased risk for toxicity by participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events grade ≥ 3 as assessed by CTCAEv5 | 24 hours

SECONDARY OUTCOMES:
Occurrence of adverse events grade ≥ 3 as assessed by CTCAEv5 | 100 days
Severity and duration of grade ≥ 3 mucosal toxicities including oropharyngeal mucositis, nausea, vomiting, and/or diarrhea. | Day 0 to hospital discharge
Time to neutrophil engraftment | First of three consecutive days after ASCT of absolute neutrophil count (ANC) > 500/μL
Time to platelet engraftment | First of seven consecutive days after ASCT of platelet count ≥ 20,000/μL without transfusion support
Time to lymphoid recovery | 14, 28 and 100 days post-ASCT
Progression-free survival | 100 and 365 days post-ASCT
Non-relapse mortality | 100 and 365 days post-ASCT
Overall survival | 100 and 365 days post-ASCT

CONTACTS AND LOCATIONS:
Overall Officials: Paul Finnegan, MD, Study Director — Angiocrine Bioscience
Locations (9):
- United States (9):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - UC San Diego Moores Cancer Center, San Diego, California
  - The University of California San Francisco, San Francisco, California
  - University of Michigan, Ann Arbor, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson, Houston, Texas

IPD SHARING:
Plan to Share IPD: No